CLINICAL TRIAL: NCT02473198
Title: A Prospective Randomized Trial Comparing Femoral Nerve Black to Intraoperative Local Anesthetic Injection of Liposomal Bupivacaine (Exparel) in Total Knee Replacement
Brief Title: Femoral Nerve Block Compared to Exparel in Total Knee Replacement
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The New England Baptist Hospital (Other)
Responsible Party: Principal Investigator, Carl Talmo, Principal Investigator, The New England Baptist Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 463360
Record Dates: First submitted 2015-01-05; First posted 2015-06-16 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-03

CONDITIONS: Osteoarthritis; Pain
Keywords: Total Knee Arthroplasty; Amide Local Anesthetic
MeSH Terms: conditions — Osteoarthritis; Pain | interventions — Bupivacaine; Ketorolac Tromethamine; Ketorolac; Morphine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Femoral Nerve Block (Group 1) (Active Comparator): In group1 (standard group) all patients receive the standard current perioperative pain management protocol for TKR.
  The patient will then undergo an ultrasound guided femoral nerve block with bupivacaine 0.25% 20 cc. Intraoperatively prior to cementing of the TKR, patients will also receive a local anesthetic injection of a mixture of 30cc 0.25% bupivicaine with epinephrine, 30mg of toradol and 10 mg of morphine sulfate into the posterior capsule of the knee joint. Postoperatively patients will receive narcotic pain medication on a PRN basis.
  Interventions: Drug: Femoral Nerve Block Bupivacaine
- Exparel (Group 2) (Experimental): Group 2 will receive standard perioperative pain management for TKR; will undergo placebo femoral nerve block under ultrasound guidance with normal saline (NS) 20 cc. Following femoral bone cuts they will receive local anesthetic injection mixture of 30cc 0.25% bupivicaine with epinephrine 20 cc of preservative free normal saline, 30mg of toradol and 10 mg of morphine sulfate into the periarticular tissues including periosteum, joint capsule and posterior capsule of the knee joint and collateral ligaments and subcutaneous tissues. Prior to cementing prosthesis, a second injection with mixture of 20mL 1.3% Exparel and 40mL normal saline solution will be injected into the same tissues, joint capsules and collateral ligaments.
  Interventions: Drug: Exparel; Drug: Toradol; Drug: Morphine Sulfate

INTERVENTIONS:
Drug: Exparel — Prior to cementing of the prosthesis (minimum 20 minutes later), injection with mixture of 40 mL normal saline solution and 20mL 1.3% Exparel.
  Other Names: Bupivacaine liposome injectable suspension
  Arms: Exparel (Group 2)
Drug: Femoral Nerve Block Bupivacaine — The patient will then undergo an ultrasound guided femoral nerve block in the preoperative area with bupivacaine 0.25% 20 cc. All patients will undergo unilateral TKR using a medial parapatellar approach. Intraoperatively prior to cementing of the TKR, patients will also receive a local anesthetic injection of a mixture of 30cc 0.25% bupivicaine with epinephrine, 30mg of toradol and 10 mg of morphine sulfate into the posterior capsule of the knee joint.
  Other Names: Bupivacaine
  Arms: Femoral Nerve Block (Group 1)
Drug: Toradol — The patient will then undergo an ultrasound guided femoral nerve block in the preoperative area with bupivacaine 0.25% 20 cc. All patients will undergo unilateral TKR using a medial parapatellar approach. Intraoperatively prior to cementing of the TKR, patients will also receive a local anesthetic injection of a mixture of 30cc 0.25% bupivicaine with epinephrine, 30mg of toradol and 10 mg of morphine sulfate into the posterior capsule of the knee joint.
  Other Names: Sprix; Acuvail; Acular
  Arms: Exparel (Group 2)
Drug: Morphine Sulfate — The patient will then undergo an ultrasound guided femoral nerve block in the preoperative area with bupivacaine 0.25% 20 cc. All patients will undergo unilateral TKR using a medial parapatellar approach. Intraoperatively prior to cementing of the TKR, patients will also receive a local anesthetic injection of a mixture of 30cc 0.25% bupivicaine with epinephrine, 30mg of toradol and 10 mg of morphine sulfate into the posterior capsule of the knee joint.
  Other Names: Astramorph PF; Duramorph; Infumorph
  Arms: Exparel (Group 2)

SUMMARY:
The main objective of the study is to determine if intrarticular injection with liposomal bupivicaine (Exparel) provides better postoperative pain relief and functional outcome following total knee replacement (TKR) than the current standard New England Baptist Hospital regimen of femoral nerve block combined with intraarticular injection of a standard bupivicaine solution.

DETAILED DESCRIPTION:
A prospective, single blind study comparing femoral nerve blockade and intraarticular posterior capsular injection to interarticular injection of bupivicaine and liposomal bupivicaine (Exparel) alone.

ELIGIBILITY:
Inclusion Criteria:

• Patients between the ages of 18 - 73 who are undergoing primary, unilateral, Total Knee Replacement at the New England Baptist Hospital in Boston, Massachusetts are eligible to participate.

Exclusion Criteria:

* Patients with Revision or Complex Total Knee Replacements and are under the age of 18, or over the age of 73 will be excluded.
* Patients with an ASA 4 level will be excluded.
* Patients with a Body Mass Index of less than 20, and over 40, will be excluded.
* Patients taking preoperative narcotics, patients with extreme sensitivity or allergy to narcotics or local anesthetics, and patients using opioid medications for at least 3 months leading up to surgery, will also be excluded.

Ages: 18 Years to 73 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Estimated)
Dates: Start 2014-01; Primary Completion 2017-02 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Pain Relief measured by VAS Questionnaire | One Year
  The main objective of the study is to determine if intrarticular injection with liposomal bupivicaine (Exparel) provides better postoperative pain relief and functional outcomes following total knee replacement (TKR) than the current standard NEBH regimen of femoral nerve block combined with intraarticular injection of a standard bupivicaine solution.

SECONDARY OUTCOMES:
Functional Ability measured by the KSS Questionnaire Score | One Year
  The main objective of the study is to determine if intrarticular injection with liposomal bupivicaine (Exparel) provides better postoperative pain relief and functional outcomes following total knee replacement (TKR) than the current standard NEBH regimen of femoral nerve block combined with intraarticular injection of a standard bupivicaine solution.

CONTACTS AND LOCATIONS:
Overall Officials: Carl Talmo, MD, Principal Investigator — New England Baptist Hospital
Locations (1):
- New England Baptist Hospital, Boston, Massachusetts, United States